CLINICAL TRIAL: NCT01743235
Title: A Double-blind, Randomized, Placebo-controlled, Dose-finding Study to Investigate the Safety and Efficacy of Lybridos in the Domestic Setting in Healthy Female Subjects With Hypoactive Sexual Desire Disorder and Maladaptive Activity of Sexual Inhibitory Mechanisms
Brief Title: Lybridos in Pre- and Postmenopausal Women With Hypoactive Sexual Desire Disorder Due to Maladaptive Activation of Sexual Inhibitory Systems
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emotional Brain NY Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EB90; EB90 (Other: Emotional Brain NY Inc.)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: HSDD
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Testosterone; Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Experimental): 30 subjects administered a placebo
  Interventions: Drug: Placebo
- Testosterone + Buspirone hydrochloride combination drug (Experimental): 30 subjects are given combination drug (0.25 mg Testosterone + 5 mg Buspirone hydrochloride)
  Interventions: Drug: Testosterone; Drug: Buspirone hydrochloride
- Testosterone + Buspirone hydrochloride combinat (Experimental): 30 subjects are given combination drug (0.25 mg Testosterone + 10 mg Buspirone hydrochloride)
  Interventions: Drug: Testosterone; Drug: Buspirone hydrochloride
- Testosterone + Buspirone Combination Drug (Experimental): 30 subjects are given combination drug (0.5 mg Testosterone + 5 mg Buspirone hydrochloride)
  Interventions: Drug: Testosterone; Drug: Buspirone hydrochloride
- Testosterone +Buspirone Combination Drug (Experimental): 30 subjects are given combination drug (0.5 mg Testosterone + 10 mg Buspirone hydrochloride)
  Interventions: Drug: Testosterone; Drug: Buspirone hydrochloride
- Testosterone (Experimental): 30 subjects are given 0.5 mg Testosterone
  Interventions: Drug: Testosterone
- Buspirone (Experimental): 30 subjects are given 10 mg Buspirone hydrochloride
  Interventions: Drug: Buspirone hydrochloride

INTERVENTIONS:
Drug: Placebo — Solid Oral Dosage. Maximum every other day (on an as needed basis)
  Arms: Placebo
Drug: Testosterone — Solid Oral Dosage. Maximum every other day (on an as needed basis)
  Arms: Testosterone; Testosterone + Buspirone Combination Drug; Testosterone + Buspirone hydrochloride combinat; Testosterone + Buspirone hydrochloride combination drug; Testosterone +Buspirone Combination Drug
Drug: Buspirone hydrochloride — Solid Oral Dosage. Maximum every other day (on an as needed basis)
  Arms: Buspirone; Testosterone + Buspirone Combination Drug; Testosterone + Buspirone hydrochloride combinat; Testosterone + Buspirone hydrochloride combination drug; Testosterone +Buspirone Combination Drug

SUMMARY:
A double-blind, randomized, placebo-controlled, dose-finding study to investigate the safety and efficacy of Lybridos in the domestic setting in healthy female subjects with hypoactive sexual desire disorder and maladaptive activity of sexual inhibitory mechanisms.

In the present study, the efficacy of Lybridos will be evaluated in the domestic setting in healthy female subjects with HSDD and maladaptive activity of sexual inhibitory mechanism(s). Sexual satisfaction and other aspects of sexual functioning will be measured within 24 hours after each sexual activity. The following hypotheses will be tested:

Lybridos, as compared to placebo, will significantly increase the number of satisfying sexual events.

The number of satisfying sexual events will not differ significantly between subjects treated with placebo and subjects treated with 0.5 mg testosterone alone and/or 10 mg buspirone alone.

Lybridos, as compared to placebo, will significantly increase sexual desire/arousal.

Sexual desire/arousal will not differ significantly between subjects treated with placebo and subjects treated with 0.5 mg testosterone alone and/or 10 mg buspirone alone.

Lybridos, as compared to testosterone alone and buspirone alone, will significantly increase the number of satisfying sexual events and sexual desire/arousal.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Provision of written informed consent
2. Females between 21 and 70 years of age, inclusive, pre- or postmenopausal, with HSDD (comorbidity with female sexual arousal disorder [FSAD] and/or female orgasmic disorder [FOD; only as secondary diagnosis] is allowed). The diagnosis of HSDD will be established by a trained health care professional.
3. Maladaptive activity of sexual inhibitory mechanism(s) (see appendix 5 for definition)
4. Be involved in a stable relationship and have a partner who will be accessible for the majority of the study duration
5. Healthy with normal medical history, physical examination, laboratory values, and vital signs; exceptions may be made if the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible to participate in the study:

Cardiovascular Conditions

1. Any underlying cardiovascular condition, including unstable angina pectoris, that would preclude sexual activity
2. Systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg. For subjects ≥ 60 years old and without diabetes mellitus, familial hypercholesterolemia, or cardiovascular disease: systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 90 mmHg
3. Systolic blood pressure ≤ 90 mmHg and/or diastolic blood pressure ≤ 50 mmHg. Gynecological and Obstetric Conditions
4. Use of any contraceptive containing antiandrogens (e.g. Cyproteron acetate) or(anti)androgenic progestogens (drospirenone, dienogest, chlormadinone acetate and norgestrel)
5. Use of any contraceptive or hormone replacement therapy (HRT) containing more than 50 μg/day of estrogen
6. Positive test result for Chlamydia or gonorrhea
7. Pregnancy or intention to become pregnant during this study (Note: A urine pregnancy test will be performed in all women of child bearing potential prior to the administration of study medications.)
8. Lactating or delivery in the previous 6 months prior to signing Informed Consent Form
9. Significant abnormal Pap smear in the previous 12 months prior to signing Informed Consent Form
10. History of bilateral oophorectomy
11. Other unexplained gynecological complaints, such as clinically relevant abnormal uterine bleeding patterns
12. Perimenopausal status (cycle shortening/irregular menstrual bleeding in the last 12 consecutive months and/or occurrence of vasomotor symptoms (e.g. hot flashes, night sweating) in combination with elevated FSH levels (>40 IU/L) for women from age 40 onwards; in women with a history of hysterectomy, perimenopausality can be assessed by FSH levels (> 40 IU/L) and/or vasomotor symptoms) Other Medical Conditions
13. Liver and/or renal insufficiency (aspartate aminotransferase, alanine aminotransferase and gamma glutamyltransferase > 3 times the upper limit of normal and/or estimated glomerular filtration rate (eGFR) < 60.00 mL/min based on the Cockcroft-Gault formula)
14. Any current endocrine disease or endocrinopathy (e.g. uncontrolled thyroid dysfunction) as determined by medical history, basic physical examination and/or laboratory values significantly outside normal range of the central laboratory; or uncontrolled diabetes mellitus (HbA1c > 7.5%)
15. Free- and/or total testosterone levels outside the upper limit of the reference range of the central laboratory (free testosterone: > 1.1 ng/dL, and total testosterone > 80 ng/dL)
16. Any current clinically relevant neurological disease which, in the opinion of the investigator, would compromise the validity of study results or which exclude from use of buspirone and/or testosterone
17. History of hormone-dependent malignancy (including all types of breast cancer)
18. Vision impairment, such as partial or complete blindness or color blindness
19. Dyslexia
20. Positive test result for immunodeficiency virus, hepatitis B, or hepatitis C (acute and chronic hepatitis infection)
21. History of serotonin syndrome Psychological/Psychiatric Factors
22. History of (childhood) sexual abuse that, in the opinion of the investigator, could result in negative psychological effects when testosterone is administered
23. (Psychotherapeutic and/or pharmacological treatment for) a psychiatric disorder that, in the opinion of the investigator, would compromise the validity of study results or which could be a contraindication for buspirone and/or testosterone use
24. Current psychotherapeutic treatment for female sexual dysfunction
25. Current sexual disorder of vaginismus or dyspareunia according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (text revision (DSM-IV-TR))
26. A substance abuse disorder that, in the opinion of the investigator, is likely to affect the subject's ability to complete the study or precludes the subject"s participation in the study (mild or moderate alcohol consumption is allowed but must be stopped 12 hours before the Stroop task).
27. A score of > 65 at the STAI-Y2 questionnaire
28. Positive test result for illicit drugs Concomitant Medications
29. Use of potent CYP3A4 inhibitors (eg, ritonavir, ketoconazole, itraconazole clarithromycin, erythromycin and saquinavir)
30. Use of potent CYP3A4 inducers (eg, carbamazepine, phenytoin, phenobarbital, St John"s wort, rifampin)
31. Use of selective serotonin reuptake inhibitors, tricyclic antidepressants or other antidepressants
32. Use of any other medication that interferes with study medication (eg, monoamine oxidase [MAO] inhibitors [includes classic MAO inhibitors and linezolid],spironolactone)
33. Use of medication (including herbs) that would compromise the validity of study results
34. Use of testosterone therapy within 6 months before study entry prior to signing the Informed Consent Form General
35. Illiteracy, unwillingness, or inability to follow study procedures
36. Participation in other clinical trials within the last 30 days
37. Any other clinically significant abnormality or condition which, in the opinion of the investigator, might interfere with the participant"s ability to provide informed consent or comply with study instructions, compromise the validity of study results, or be a contraindication for buspirone and/or testosterone use

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Satisfactory Sexual Episodes | 20 Weeks
  To investigate the efficacy of Lybridos as compared to placebo in increasing the number of satisfactory sexual episodes in healthy female subjects with hypoactive sexual desire disorder(HSDD) and maladaptive activity of sexual inhibitory mechanisms

SECONDARY OUTCOMES:
Sexual satisfaction | 20 Weeks
  Sexual satisfaction will be evaluated based on a global satisfaction assessment comparing the 4-week establishment period with the 8 week DB treatment period. In addition there is a 8 week run in period between the establishment period and the double blind treatment period for a total treatment period of 20 weeks.
Sexual desire and arousal | 20 Weeks
  Sexual desire and arousal will be evaluated based on the 'desire' and 'arousal' domains of the Sexual Anamnesis Questionnaire, the Sexual Function questionnaire and weekly diaries throughout the course of the study.
Sexual motivation and inhibition | 20 weeks
  Sexual motivation and inhibition will be assessed using the Sexual Motivation Questionnaire and comparing sexual motivation and inhibition between the 4-week establishment period and the 8-week DB treatment period. In addition there is a 8 week run in period between the establishment period and the double blind treatment period for a total treatment period of 20 weeks.
Safety and toleration | 20 weeks
  Safety will be evaluated by: 1) AEs [Number of patients reporting AEs, number of patients reporting drug related AEs] 2)SAE [Number of patients reporting SAEs, number of patients reporting drug related SAEs]and 3) Changes in laboratory safety data [Number of patients reporting abnormal lab safety data, number of patients reporting drug related abnormal lab safety data]. These will be evaluated throughout the course of the study.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - San Diego Sexual Medicine, San Diego, California
  - Meridien Research, Bradenton, Florida
  - Segal Insitute for Clinical Research, North Miami, Florida
  - Compass Research, Orlando, Florida
  - Meridien Research, St. Petersburg, Florida
  - Annapolis Sexual Wellness Center, Annapolis, Maryland
  - Maryland Prime Care Physicians, Stevensville, Maryland
  - Center for Sexual Medicine at Sheppard Pratt, Townson, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - NECCR Fall River LLC, Fall River, Massachusetts
  - Michael A. Werner, MD PC, Purchase, New York
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania